CLINICAL TRIAL: NCT03998085
Title: Study of Anlotinib Single Drug as the Maintenance Treatment for Advanced Non-Small Cell Lung Cancer （NSCLC）
Brief Title: Anlotinib Single Drug as the Maintenance Treatment for Advanced NSCLC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Hospital of Jilin University (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K2018065; ALTER-L011 (Other: Chia Tai Tianqing Pharmaceutical Group Co., Ltd.)
Record Dates: First submitted 2019-06-23; First posted 2019-06-25 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anlotinib (Experimental)
  Interventions: Drug: Anlotinib Hydrochloride

INTERVENTIONS:
Drug: Anlotinib Hydrochloride — Anlotinib hydrochloride capsule 12 mg, orally, once a day, oral before breakfast, according to the research program for 2 weeks, discontinued for 1 week. Patients with complete remission (CR), partial remission (PR) and stable disease (SD) continued to administer drugs until the disease progressed, intolerable toxicity or withdrawal was required. Patients with progression of illness (PD) discontinued their medication.

SUMMARY:
Based on the need of clinical practice of maintenance therapy for advanced NSCLC and the reliable data of third-line treatment for non-small cell lung cancer, the investigators designed a clinical study of anlotinib in maintenance therapy for advanced NSCLC to prospectively evaluate the efficacy of anlotinib in maintenance therapy for advanced NSCLC. Value, to provide a scientific basis for prolonging the survival time of patients with advanced NSCLC, improving the quality of life of patients in the course of treatment, and optimizing treatment strategies to a greater extent.

ELIGIBILITY:
Inclusion Criteria:

* a.NSCLC was diagnosed by cytology or histology, and patients with stage IIIB,IIIC or IV and no sensitive mutation of EGFR/ALK were diagnosed according to UICC Staging Standard of the 8th edition of 2017; b. Patients with disease recurrence or progression 1 year after radical operation with platinum-assisted chemotherapy;
* Those who had received platinum-containing two-drug combination chemotherapy for 4-6 cycles were judged as complete remission (CR), partial remission (PR) and stabilization (SD) according to RECIST 1.1 standard;
* Patients should be enrolled after the end of the last first-line chemotherapy cycle with platinum containing drugs ≤6 weeks (42 days)
* Age: 18 to 75 years old
* PS<2(ECOG) ;
* The life expectancy is more than 3 months;
* According to RECIST 1.1 criteria, patients have at least one imaging (CT, MRI) lesion that can be measured or evaluated; the lesion was not previously treated by radiotherapy. The longest diameter of the target lesion should be greater than or equal to 10 mm (the short axis of lymph node is greater than or equal to 15 mm); Patients with brain metastasis at baseline should be single intracranial metastasis, asymptomatic or asymptomatic after treatment;
* Women: For all women who may be pregnant, pregnancy tests must be performed within 72 hours before starting treatment, or medically approved contraceptive methods must be used within three months after the treatment and during the period after the end of treatment; serum or urine pregnancy tests must be negative and must be non-lactating; Male: Contraceptive measures were taken during and within 3 months after surgical sterilization or treatment;
* The functional level of organs must meet the following requirements:

Routine blood test ANC≥1.5 x 109/L; PLT≥100 x 109/L; Hb≥90g/L Blood biochemistry TBIL≤1.5 x ULN ALT and AST≤2 x ULN; for patients with liver metastases, ALT and AST ≤5 x ULN; BUN and Cr≤1.5 x ULN and creatinine clearance≥50 ml/min；LVEF≥50%; 12 lead electrocardiogram The Fridericia-corrected QTcF was < 450 ms for males and < 470 MS for females.

* Subjects who have the ability to understand and sign the informed consent must sign the informed consent before any screening evaluation.

Exclusion Criteria:

* Small cell lung cancer (including mixed small cell lung cancer and non-small cell lung cancer);Central squamous cell carcinoma, or non-small cell lung cancer with hemoptysis (> 50ml/d) or risk of massive bleeding;
* Imaging (CT or MRI) shows that the distance between tumor lesion and the large blood vessel is ≤ 5 mm, or there is a central tumor that invades the local large blood vessel; or there is a significant pulmonary cavity or necrotizing tumor;
* Medical history and combined history

  1. Active brain metastases, cancerous meningitis, spinal cord compression, or imaging CT or MRI screening for brain or pia mater disease;
  2. The patient is participating in other clinical studies or completing the previous clinical study in less than 4 weeks;
  3. Patients with hypertension who could not be well controlled by antihypertensive drug (systolic pressure > 150 mmHg, diastolic pressure > 100 mmHg);
  4. Had malignant tumors except NSCLC within 5 years before enrollment(except for patients with cervical carcinoma in situ , basal cell or squamous cell skin cancer who have undergone a curative treatment, local prostate cancer after radical resection, ductal carcinoma in situ or papillary thyroid cancer after radical resection);
  5. Researchers judged that they had not recovered from previous adverse events before taking the drug for the first time (NCI-CTCAE Version 4.0 Grade > Grade 1);
  6. Abnormal blood coagulation (INR > 1.5 or prothrombin time (PT) > ULN + 4 seconds or APTT > 1.5 ULN), with bleeding tendency or undergoing thrombolytic or anticoagulant therapy;Note: Under the premise of prothrombin time international normalized ratio (INR) ≤ 1.5, low-dose heparin (adult daily dose of 0.6 million to 12,000 U) or low-dose aspirin (daily dosage ≤ 100 mg) is allowed for preventive purposes;
  7. Renal insufficiency: urine routine indicates urinary protein ≥ ++, or confirmed 24-hour urine protein ≥ 1.0g;
  8. The effects of surgery or trauma have been eliminated for less than 14 days before enrollment in subjects who have undergone major surgery or have severe trauma;
  9. Severe acute or chronic infections requiring systemic treatment;
  10. Suffering from severe cardiovascular disease: myocardial ischemia or myocardial infarction above grade II, poorly controlled arrhythmias (including men with QTc interval ≥ 450 ms, women ≥ 470 ms); according to NYHA criteria, grades III to IV Insufficient function, or cardiac color Doppler ultrasound examination indicates left ventricular ejection fraction (LVEF) <50%;
  11. There is currently a peripheral neuropathy of ≥CTCAE 2 degrees, except for trauma;
  12. Respiratory syndrome (≥CTC AE grade 2 dyspnea), serous effusion (including pleural effusion, ascites, pericardial effusion) requiring surgical treatment;
  13. There was a history of bleeding. Within 4 weeks before screening, any bleeding events with a severe grade of 3 or more in CTCAE 4.0 occurred;
  14. Decompensated diabetes or other ailments treated with high doses of glucocorticoids;
  15. Factors that have a significant impact on oral drug absorption, such as inability to swallow, chronic diarrhea, and intestinal obstruction;
  16. Clinically significant hemoptysis (daily hemoptysis greater than 50ml) within 3 months prior to enrollment; or significant clinically significant bleeding symptoms or defined bleeding tendency, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, baseline fecal occult blood ++ and above, or suffering from vasculitis;
  17. Events of venous/venous thrombosis occurring within the first 6 months prior to enrollment, such as cerebrovascular accidents (including transient ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism;
  18. Participated in clinical trials of other anti-tumor drugs during the first 4 weeks of enrollment or planned systemic anti-tumor therapy, including cytotoxic therapy, signal transduction inhibitors, immunotherapy (or mitomycin C during the first 6 weeks of trial drug treatment), or during the first 4 weeks of study administration.In the first 4 weeks of the study, the patients were treated with ef-rt or field-limited radiotherapy for tumor lesion evaluation.
  19. Those with allergic constitution or known history of allergy to the drug components of this regimen;
  20. Has a history of immunodeficiency, including HIV positive testing, or other acquired, congenital immunodeficiency disorders, or organ transplantation history;
  21. The baseline pregnancy test was positive for pregnant, lactating or fertile women, and the patients of childbearing age who were unwilling to take effective contraceptive measures during the whole period of the test were unwilling to take effective contraceptive measures;
  22. According to the judgement of researchers, there are concomitant diseases that seriously endanger patients'safety or affect patients' completion of research;
  23. There was a clear history of neurological or psychiatric disorders, including epilepsy or dementia;
  24. Cirrhosis, decompensated liver disease, untreated active hepatitis(HBV: HBsAg positive and DNA≥500IU/Ml;HCV:RNA positive and abnormal liver function);Co-infection with HBV and HCV;
  25. Renal failure requires hemodialysis or peritoneal dialysis.
* According to the researcher's judgment, the patient may have other factors that may lead to the forced termination of the study, such as other serious diseases or serious laboratory abnormalities or other factors that may affect the safety of the subjects, or family or social factors that may affect the collection of test data and samples

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-03-05 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | 5 months
  Progression free survival

SECONDARY OUTCOMES:
OS | through study completion, an average of 18 months
  Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No